CLINICAL TRIAL: NCT05675956
Title: Exploration of Acute Nerve Stimulation by Way of Novel ApolloNeuro™ Device and Its Influences on Physiological Function to Mediate Human Performance and Cognition
Brief Title: Acute Nerve Stimulation For Enhancing Human and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00122153
Record Dates: First submitted 2022-11-02; First posted 2023-01-09 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Concussion, Mild; Autonomic Nervous System; Cognitive
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Participants will participate in both arms of the intervention.
Who Masked: Participant
Masking Description: This will be a single-blind study, the investigators will know which condition subjects are assigned at which visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity (Experimental): The device will be set to 100% intensity for this group.
  Interventions: Device: Experimental group with 100% intensity setting on Apollo Neuro device
- Low Intensity (Active Comparator): The device will be set to 10% intensity in this group
  Interventions: Device: Active Comparator group with 10% intensity setting on the Apollo Neuro device

INTERVENTIONS:
Device: Experimental group with 100% intensity setting on Apollo Neuro device — The group will have the device set to 100% intensity at one of their two experimental visits.
  Arms: High Intensity
Device: Active Comparator group with 10% intensity setting on the Apollo Neuro device — The group will have the device set to 10% intensity at one of their two experimental visits.
  Arms: Low Intensity

SUMMARY:
The goal of this clinical trial is to test a wearable device's effect on performance in tactical populations with a history of concussion. The main question it aims to answer is the effectiveness of the device on modulate physiological and cognitive function.

The physiological function will be derived from metrics of heart rate variability and blood-based biomarkers, whilst human performance will be evaluated using tasks that assess cognitive domains of executive function, reaction time, and memory.

DETAILED DESCRIPTION:
This study will compare the effects of two different settings of the ApolloNeuro™ Device on physiological and cognitive function. This device is worn on the wrist and produces silent low-frequency waves that feel like slight vibrations. The purpose of the device is to modulate autonomic nervous system function. There will be a total of 3 laboratory visits, each lasting approximately 3.5 hours, separated by 3-5 days to allow for physiological recovery. The first visit will include an exercise test to determine participants maximum exercise capacity and to familiarize participants with a battery of psycho-motor cognitive tasks. The remaining two visits will be experimental days differentiated by a low or high-intensity setting of the ApolloNeuro™ Device. The experimental order will be randomized. This means that neither the participant nor the research team will know which condition has been assigned. On the experimental days, participants will have blood drawn from their arm and complete psycho-motor cognitive measures before and after a 20-minute interval running workout. This study will help to acquire knowledge of how wearable devices may improve physiological and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between 18-30 BMI.
* Participant needs to be either an ROTC member, currently employed military or law enforcement officer or are a military veteran or retired law enforcement officer who has completed service in the past 18 months.
* Participant has provided written and dated informed consent.
* Participant is in good health and able to participate in high-intensity exercise.
* Participant have been clinically diagnosed with a concussion at least 3 months prior to screening and is asymptomatic.
* Participant is willing to maintain their current dietary supplement usage through the duration of the study. If the participant began taking another supplement within the past month, the participant will be asked to discontinue supplement use followed by a 2-week washout prior to participation.

Exclusion Criteria:

* Participant with any musculoskeletal injuries that would prevent exercising.
* Participant with any metabolic disorder including known electrolyte abnormalities, diabetes, thyroid disease, adrenal disease or hypogonadism.
* Participant with a history of hepatorenal, musculoskeletal, or autoimmune disease.
* Participant with a personal history of heart disease, cardiovascular conditions, high blood pressure (systolic >140 mm Hg & diastolic >90 mm Hg), psychiatric disorders, neurological disorders, developmental disorders, cancer, benign prostate hypertrophy, gastric ulcer, reflux disease, or any other medical condition (i.e. visual/auditory) deemed exclusionary by the medical staff.
* Participant currently taking medication that affects the ANS such as thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, anticoagulant, or psychotropic medications, or antihistamines.
* Participant who is pregnant or lactating.
* Participant with any of the following concussion characteristics; history of >3 concussions, loss of consciousness (>5 minutes), cause of injury related to violence e.g. physical altercations.
* Participants with a history of moderate to severe TBI.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Changes in dopamine | Will be assessed at visits 2 and 3 prior exercise (minute 0) , immediately following exercise (about 1.5 hour), and immediately post one hour recovery (at about hour 3) on experimental visits.
  To determine if the device has an impact on dopamine levels
Changes in epinephrine | Will be assessed at visits 2 and 3 prior exercise (minute 0) , immediately following exercise (about 1.5 hour), and immediately post one hour recovery (at about hour 3) on experimental visits.
  To determine if the device has an impact on epinephrine levels
Changes in norepinephrine | Will be assessed at visits 2 and 3 prior exercise (minute 0) , immediately following exercise (about 1.5 hour), and immediately post one hour recovery (at about hour 3) on experimental visits.
  To determine if the device has an impact on norepinephrine levels
Changes in cortisol | Will be assessed at visits 2 and 3 prior exercise (minute 0) , immediately following exercise (about 1.5 hour), and immediately post one hour recovery (at about hour 3) on experimental visits.
  To determine if the device has an impact on cortisol levels
Changes in arousal | Will be assessed at visits 2 and 3 prior exercise (minute 0) on experimental visits.
  To determine if the device has an impact on arousal levels measured by the "Felt Arousal Scale". The minimum score is 1 and maximum score is 6. These measures are not indicative of better or worse outcomes.
Sleep Quality | Will be assessed at visits 2 and 3 prior exercise (minute 0) on experimental visits.
  Index of sleep quality using the Neurology Quality of Life (Neuro-QOL) sleep subscale.
Changes in fatigue | Will be assessed prior exercise (minute 0), immediately after the bout of exercise (about hour 1.5), post cognitive testing (about 2 hour), and immediately post one hour recovery (about hour 3) on experimental visits.
  To determine if the device has an impact on fatigue levels measured by the "Fatigue Scale". The minimum score is 1 and maximum score is 5. These measures are not indicative of better or worse outcomes.
Changes in Marksmanship Accuracy | Will be assessed prior exercise (minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  Simulated marksmanship using optical targetry
Changes in Marksmanship Reaction Time | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  Simulated marksmanship using optical targetry
Changes in cognitive flexibility by local switch cost RT (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive flexibility by measuring local switch cost RT within the heterogenous condition when switching rule sets represented as the additional time to respond to switch relative to repeat trials.
Changes in cognitive flexibility by local switch cost ACC (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive flexibility by measuring local switch cost ACC within the heterogenous condition when switching rule sets represented as the difference between error rates for switch relative to repeat trials.
Changes in cognitive flexibility by local switch cost IES (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive flexibility by measuring local switch cost inverse efficiency scores (IES) represented as dividing RTs by 1 minus the percentage of errors (i.e., percentage of correct responses).
Changes in global executive function by global cost RT (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on global executive function by measuring global cost RT represented as the difference between the time required to respond between the heterogeneous and homogeneous conditions.
Changes in global executive function by global cost ACC (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on global executive function by measuring global cost ACC represented as the difference between error rates between homogeneous and heterogeneous conditions.
Changes in global executive function by global cost IES (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on global executive function by measuring global cost IES.
Changes in working memory by mixing cost RT (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on working memory by measuring mixing cost RT represented as the additional time required to respond between the repeat trials in the heterogenous condition relative to the trials in the homogeneous condition.
Changes in working memory by mixing cost ACC (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on working memory by measuring mixing cost ACC represented as the difference in error rates on repeat trials in the heterogenous condition relative to the trials in the homogeneous condition.
Changes in working memory by mixing cost IES (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on working memory by measuring mixing cost IES.
Changes in attention (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention measured by the omission errors when an individual fails to respond to a color-switch task trial, and omission error runs when an individual fails to respond to multiple successive trials.
Changes in Inhibitory Control (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on inhibitory control measured by the commission errors when an individual fails to respond correctly to a color-switch task trial, and commission error runs when an individual fails to respond correctly to multiple successive trials.
Changes in attention and cognitive control by ACC (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention and cognitive control by measuring heterogeneous condition ACC.
Changes in attention and cognitive control by RT (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention and cognitive control by measuring heterogeneous condition RT.
Changes in attention and cognitive control by IES (Switch Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention and cognitive control by measuring heterogeneous condition IES.
Changes in Inhibitory Control (Go/No go) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on inhibitory control by measuring reaction time to Go targets (hits).
  To determine if the device has an impact on inhibitory control by measuring errors of commission representing incorrect responses to the target NoGo (false alarm).
Changes in Attention (Go/No go) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention by measuring errors of omission to the target Go (misses).
Changes in Autonomic Nervous System Function (ANS) by linear metrics | This will be continuously assessed throughout the entirety of experimental visits 2 and 3 (minute 0 to about 3 hours)..
  To determine if the device has an impact on ANS function by measuring heart rate variability represented by linear (RMSSD, SDNN, CVNN) time domain metrics.
Changes in Autonomic Nervous System Function (ANS) by nonlinear metrics | This will be continuously assessed throughout the entirety of experimental visits 2 and 3 (minute 0 to about 3 hours)..
  To determine if the device has an impact on ANS function by measuring heart rate variability represented by nonlinear (ApSaEn) time domain metric.
Changes in Autonomic Nervous System Function (ANS) by frequency domain metrics | This will be continuously assessed throughout the entirety of experimental visits 2 and 3 (minute 0 to about 3 hours)..
  To determine if the device has an impact on ANS function by measuring heart rate variability represented by frequency domain (HF, LF, Coherence Ratio) metrics.
Changes in Inhibitory Control by accuracy scores (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on inhibitory control measured by the accuracy scores (% of correct answers) for compatible-congruent, incompatible-congruent, compatible-incongruent, and incompatible-incongruent Flanker Task trials.
Changes in Inhibitory Control by average response time (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on inhibitory control measured by the average response time to incongruent flanker task trials irrespective of compatible or incompatible rule sets.
Changes in Inhibitory Control by commission errors (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on inhibitory control measured by the commission errors when an individual fails to respond correctly to a flanker task trial, and commission error runs when an individual fails to respond correctly to multiple successive trials.
Changes in Attention by accuracy (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention measured by the accuracy scores for congruent-compatible Flanker task trials.
Changes in Attention by average response time (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention measured by the overall average response time (milliseconds) to compatible and incompatible Flanker task trails irrespective of trial congruency.
Changes in Attention by omission errors (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attention measured by the omission errors when an individual fails to respond to a flanker task trial, and omission error runs when an individual fails to respond to multiple successive trials.
Changes in Cognitive flexibility by accuracy (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive flexibility by the accuracy scores for incongruent-incompatible Flanker task trials.
Changes in Cognitive flexibility by average response time (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive flexibility measured by the average response time to incongruent-incompatible flanker task trials.
Changes in Cognitive control by post-error accuracy (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive control measured by post-error accuracy on Flanker task trials following an error.
Changes in Cognitive control by sequential congruency effect (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine changes in cognitive control measured by sequential congruency effect when lower interference occurs following an incongruent relative to a congruent flanker task trial reflecting a consciously controlled narrowing of attention to the central target.
Changes in Cognitive control by inverse efficiency (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on cognitive control measured by inverse efficiency a metric of a speed-accuracy trade-off for Flanker task trials.
Changes in Attentional Inhibition (Flanker Task) | Will be assessed prior exercise (about minute 30) and immediately following the bout of exercise (about hour 1.5) on experimental visits.
  To determine if the device has an impact on attentional inhibition measured by congruency interference representing the costs associated with the interference demands associated with incongruent vs congruent flanker task trials.
Changes in verbal learning (HVLT) | Will be assessed prior exercise (about minute 30), immediately following the bout of exercise (about 1.5 hours), and immediately post one hour recovery (about hour 3) on experimental visits.
  To determine if the device has an impact on verbal learning by measuring total recall score via combining the word recall score from the three trials.
Changes in memory recall (HVLT) | Will be assessed prior exercise (about minute 30), immediately following the bout of exercise (about 1.5 hours), and immediately post one hour recovery (about hour 3) on experimental visits.
  To determine if the device has an impact on memory by measuring delayed recall via the delayed recall score.
Changes in retention (HVLT) | Will be assessed prior exercise (about minute 30), immediately following the bout of exercise (about 1.5 hours), and immediately post one hour recovery (about hour 3) on experimental visits.
  To determine if the device has an impact on memory by measuring retention via dividing the delayed recall trial by the score obtained on the trial prior exercise.
Changes in memory retention (HVLT) | Immediately post one hour recovery (hour 3) on experimental visits.
  To determine if the device has an impact on memory by measuring retention via calculating a retention discrimination index by subtracting the total number of false positives from the total number of true positives.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No